CLINICAL TRIAL: NCT01461239
Title: Randomized Clinical Comparison of Endodontically Treated Teeth Restored With Fiber Posts or Cast Metal Posts
Brief Title: Clinical Comparison of Endodontically Treated Teeth Restored With Fiber Posts or Cast Metal Posts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Collaborators: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Coordinator of Clinical Trials, Graduate Program in Dentistry, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFPEL-PPGO0010
Record Dates: First submitted 2011-07-05; First posted 2011-10-28 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Post and Core Failure
Keywords: survival; debonding; endodontic treated teeth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- cast post and core (Active Comparator)
  Interventions: Procedure: cast post and core
- fiber post - self-adhesive cement (Experimental)
  Interventions: Procedure: fiber post and resin core - self-adhesive cement
- fiber post - conventional cement (Experimental)
  Interventions: Procedure: fiber post luted with conventional resin cement

INTERVENTIONS:
Procedure: fiber post and resin core - self-adhesive cement — pre-fabricated glass fiber posts, cemented with self-adhesive resinous cement
  Arms: fiber post - self-adhesive cement
Procedure: cast post and core — Ni-Cr alloy cast post and core luted with self-adhesive resin cement
  Arms: cast post and core
Procedure: fiber post luted with conventional resin cement — fiber post luted with conventional etch-and-rinse adhesive system and conventional resin cement, followed by core construction with composite resin
  Arms: fiber post - conventional cement

SUMMARY:
There are few randomized controlled trials comparing intraradicular posts used to restore endodontically treated teeth, especially considering cast posts and glass fiber posts. The investigators study will evaluate the clinical success rates of endodontically treated teeth restored with glass fiber posts or cast posts and metal ceramic crown. Individuals included in this study should present any tooth with endodontic treatment and need of intraradicular retention (post) on maxilla or mandible according to inclusion and exclusion criteria. Individuals will be randomly allocated into two groups: (1) endodontically treated teeth restored with fiber post and composite resin core and metal ceramic crown or (2) endodontically treated teeth restored with cast post and core and metal ceramic crown. A sample size calculation will be performed to establish the number of posts needed for comparison. All crowns and posts will be cemented with self-adhesive cement. Individuals will be examined by calibrated examiners, in years 1 to 3. The reason of failure will be categorized as root fracture, fracture of the post, post debonding, clinical and/or radiographical evidence of a gap between restoration and tooth or endodontic failure, tooth extraction, secondary caries, or marginal defects. The confidence level will be set in 95%.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with normal occlusion with at least one teeth endodontically treated needing restoration

Exclusion Criteria:

* patients with malocclusion,
* orthodontic devices,
* temporomandibular disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Post and core survival | 72 months

SECONDARY OUTCOMES:
patient satisfaction with the treatment | 18 months
quality of crowns and restorations (FDI criteria) | 18 months
endodontic success | 18 months
  assessed by periapical radiographs for observation of apical lesion presence or absence

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Pereira-Cenci, PhD, Principal Investigator — Federal University of Pelotas; Rogério Castilho Jacinto, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- School of Dentistry - Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Bergoli CD, Machry RV, Schwantz JK, Brondani LP, Pereira-Cenci T, Pereira GKR, Valandro LF. Survival rate and treatment success of glass fiber posts cemented with two adhesive cementation strategies after up to 106 months: a randomized clinical trial. Clin Oral Investig. 2023 May;27(5):2197-2206. doi: 10.1007/s00784-023-04939-x. Epub 2023 Mar 9. PMID 36894666
- [Derived] Sarkis-Onofre R, Amaral Pinheiro H, Poletto-Neto V, Bergoli CD, Cenci MS, Pereira-Cenci T. Randomized controlled trial comparing glass fiber posts and cast metal posts. J Dent. 2020 May;96:103334. doi: 10.1016/j.jdent.2020.103334. Epub 2020 Apr 14. PMID 32302640
- [Derived] Skupien JA, Cenci MS, Opdam NJ, Kreulen CM, Huysmans MC, Pereira-Cenci T. Crown vs. composite for post-retained restorations: A randomized clinical trial. J Dent. 2016 May;48:34-9. doi: 10.1016/j.jdent.2016.03.007. Epub 2016 Mar 11. PMID 26976553